CLINICAL TRIAL: NCT02526238
Title: The Treatment Effectiveness of Theta Burst Stimulation and Voluntary Trunk Rotation for Patients With Unilateral Neglect in Stroke
Brief Title: Effectiveness of Theta Burst Stimulation (TBS) and Voluntary Trunk Rotation for Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marko Chan, Occupational Therapist, PhD Candidate, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC/KE-15-0035
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: transcranial magnetic stimulation; trunk rotation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMS and trunk rotation (Experimental): TMS and trunk rotation
  Interventions: Device: TMS and trunk rotation
- Sham TMS and trunk rotation (Sham Comparator): Sham TMS and trunk rotation
  Interventions: Device: Sham TMS and trunk rotation

INTERVENTIONS:
Device: TMS and trunk rotation — TMS and trunk rotation
  Arms: TMS and trunk rotation
Device: Sham TMS and trunk rotation — Sham TMS and trunk rotation
  Arms: Sham TMS and trunk rotation

SUMMARY:
This is a double blinded, randomized control trial with a pretest-posttest control and interventional group design. The assessor is blinded to all assessments and evaluations. All patients with subacute stroke undergo in-patient or out-patient rehabilitation are screened initially by a series of screening test. Suitable patients are assigned randomly to two groups respectively. Group 1 is the experimental group for Transcranial Magnetic Stimulation (TMS) and trunk rotation; Group 2 is the control group with only trunk rotation training and placebo stimulation.

DETAILED DESCRIPTION:
Methodology

Sampling:

Convenient sampling will be conducted to all in and out-patients with stroke referred consecutively to occupational therapy department in Kowloon Hospital during the data collection period. Patients who meet the following inclusion criteria are admitted for study.

Inclusion criteria

1. First or second stroke (haemorrhagic or ischaemic) confirmed by computer axial tomography scan or magnetic resonance imaging
2. Neurological representation compatible with a unilateral right lesion involvement (i.e. left hemiplegic), exhibited left visual field inattention or neglect by following either one of below criteria:

   * obtaining a total score of star cancellation subtest in the conventional battery of the Behavioral Inattention Test <51 (out of 54)
   * obtaining a total score of line bisection subtest in the conventional battery of the Behavioral Inattention Test <7 (out of 9)
   * Score of Catherine Bergego Scale ≥ 1
3. Right handed
4. Less than six months since onset of stroke at study entry
5. Able to follow simple command

Exclusion criteria

1. Patients with severe dysphasia (either expressive or comprehensive) which restricts communication;
2. History of other neurological disease, psychiatric disorder, or alcoholism;
3. significant impairment in visual acuity caused by cataracts, diabetic retinopathy, glaucoma or hemianopia
4. Any additional medical or psychological condition that would affect their ability to comply with the study protocol.

Data Collection and Treatment Procedures Written consent is obtained from all subjects before the randomization. All patients in both the experimental and placebo groups undergo the same rehabilitation process. Subject's demographic data are collected; they include age, gender, lesion site, educational level, time after onset of stroke, and global cognitive status as defined by the Mini-mental State Examination - Chinese version (CMMSE). Repeated measurements are done at day 0 (date for initial assessment), day 10 (end of treatment) and post 4 weeks. Assessments including Behavioral Inattention Test (BIT) - Chinese version, Catherine Bergego Scale, Functional Test for the hemiplegic upper extremity (FTHUE-HK), Upper-extremity portion of the Fugl-Meyer Scale (UE-FM), Functional Independence Measure (FIM), Stroke Adapted 30 item version of the Sickness Impact Profile (SA-SIP 30) score will be done at these intervals by a blind assessor.

Treatment sessions for the experimental groups and control groups are conducted by trained investigator for transcranial magnetic stimulation (TMS) and the case therapists. The conventional treatment would consist of 45 minutes of voluntary trunk rotation exercise using set-up equipment as well as 15 minutes of activities of daily living (ADL) training.

ELIGIBILITY:
Inclusion Criteria:

1. First or second stroke (haemorrhagic or ischaemic) confirmed by computer axial tomography scan or magnetic resonance imaging
2. Neurological representation compatible with a unilateral right lesion involvement (i.e. left hemiplegic), exhibited left visual field inattention or neglect by following either one of below criteria:

   * obtaining a total score of star cancellation subtest in the conventional battery of the Behavioural Inattention Test <51 (out of 54)
   * obtaining a total score of line bisection subtest in the conventional battery of the Behavioural Inattention Test <7 (out of 9)
   * Score of Catherine Bergego Scale ≥ 1
3. Right handed
4. Less than six months since onset of stroke at study entry
5. Able to follow simple command

Exclusion Criteria:

1. Patients with severe dysphasia (either expressive or comprehensive) which restricts communication;
2. History of other neurological disease, psychiatric disorder, or alcoholism;
3. significant impairment in visual acuity caused by cataracts, diabetic retinopathy, glaucoma or hemianopia
4. Any additional medical or psychological condition that would affect their ability to comply with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2020-03 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change score in Behaviorial Inattention Test (BIT) - Chinese version | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks), 4 weeks follow up after last session of treatment
  assessment for unilateral neglect

SECONDARY OUTCOMES:
Change score in Catherine Bergego Scale | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks), 4 weeks follow up after last session of treatment
  assessment for unilateral neglect
Change score in FTHUE-HK | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks), 4 weeks follow up after last session of treatment
  assessment for upper limb function
Change score in UE-Fugl Meyer | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks), 4 weeks follow up after last session of treatment
  assessment for upper limb function
Change score in FIM | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks time), 4 weeks follow up after last session of treatment
  assessment for activities of daily living
Change score in SA-SIP 30 | Day 0 (Date of initial assessment before treatment), Day 10 (Date after last session of treatment, expected average 3 weeks), 4 weeks follow up after last session of treatment
  assessment for well being

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yeung, MBChB, Principal Investigator — Kowloon Hospital
Locations (1):
- Kowloon Hospital, Kowloon, Hong Kong

REFERENCES:
- [Background] Fong KN, Chan MK, Ng PP, Tsang MH, Chow KK, Lau CW, Chan FS, Wong IP, Chan DY, Chan CCh. The effect of voluntary trunk rotation and half-field eye-patching for patients with unilateral neglect in stroke: a randomized controlled trial. Clin Rehabil. 2007 Aug;21(8):729-41. doi: 10.1177/0269215507076391. PMID 17846073
- [Result] Cazzoli D, Muri RM, Schumacher R, von Arx S, Chaves S, Gutbrod K, Bohlhalter S, Bauer D, Vanbellingen T, Bertschi M, Kipfer S, Rosenthal CR, Kennard C, Bassetti CL, Nyffeler T. Theta burst stimulation reduces disability during the activities of daily living in spatial neglect. Brain. 2012 Nov;135(Pt 11):3426-39. doi: 10.1093/brain/aws182. Epub 2012 Jul 24. PMID 22831781
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963